CLINICAL TRIAL: NCT04869579
Title: Selenium as a Potential Treatment for Moderately-ill, Severely-ill, and Critically-ill COVID-19 Patients
Acronym: SeCOVID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CHRISTUS Health (Other)
Collaborators: Pharco Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Mohamed Ghoweba, MD, Internal Medicine Resident Physician, CHRISTUS Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-190
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Covid19
Keywords: COVID-19 Pneumonia; Cytokine Storm; ARDS; Moderate COVID-19 Infections; Severe COVID-19 Infections; Critical COVID-19 Infections; Selenium
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — Selenious Acid

STUDY DESIGN:
Intervention Model Description: This is a randomized double-blinded, placebo-controlled Phase 2 clinical trial to assess the efficacy of Selenium in the treatment of moderately-ill, severely-ill, and critically ill COVID-19 patients. The patients will be randomized in a 1:1 ratio to receive standard of care plus a loading dose of Selenium followed by continuous infusion for a total of 14 days, or standard of care plus a Saline-based placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selenious Acid + Standard Of Care (SOC) (Experimental): Participants who are moderately-ill, severely-ill, or critically ill will receive a Selenious Acid infusion of 2000µg on day 1 as a loading dose infusion, followed by a continuous infusion of Selenious Acid at a maintenance dose of 1000µg daily on days 2-14 together with continued Standard Of Care therapy.
  Interventions: Drug: Selenium (as Selenious Acid)
- Standard Of Care (SOC) + Placebo (Active Comparator): Participants will receive a Saline-based placebo infusion of 2000µg on day 1 as a loading dose, followed by continuous infusion of a Saline-based placebo at a maintenance dose of 1000µg daily on days 2-14. Standard Of Care is to be determined according to patients' clinical picture and may include Dexamethasone, Azithromycin, Ceftriaxone, Remdesivir, Convalescent Plasma.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Selenium (as Selenious Acid) — Interventional arm participants will receive Selenium as Selenious Acid infusion plus the standard of care therapy.
  Other Names: Selenious Acid (AMERICAN REGENT)
  Arms: Selenious Acid + Standard Of Care (SOC)
Other: Placebo — Active comparator arm participants will receive the standard of care therapy plus a Saline-based placebo.
  Other Names: Saline-based Placebo
  Arms: Standard Of Care (SOC) + Placebo

SUMMARY:
Given its anti-viral, anti-oxidative, immune-enhancing, cytokine-modulating, and anticoagulant properties, the investigators hypothesize that Selenium infusion at supranutritional doses for moderately-ill, severely-ill, and critically-ill COVID-19 patients will prevent further clinical deterioration thus decreasing overall mortality and improving survival. To test this hypothesis, a prospective, single-center, phase II trial is proposed to assess the efficacy of Selenium in hospitalized adult patients with moderate, severe, and critical COVID-19 infections.

DETAILED DESCRIPTION:
COVID-19 is a respiratory illness that is caused by the novel SARS-CoV-2. Illness severity can widely range from mild, moderate, severe featuring pneumonia, to critical. Despite ongoing extensive research to find a cure for COVID-19, there had been no proven, efficacious, and widely-available treatment for the disease. With the death toll rising in various parts of the US and the world, it is imperative that investigators work on determining new therapeutic modalities. This study relates to inpatient and critical care for COVID-19 patients.

The role of Selenium (Se) as a trace element involved in many biological processes and reactions is well established in various organisms. Particularly, Selenium is known to have anti-viral, anti-oxidative, cytokine-modulating, immune-enhancing, and anticoagulant properties that might be beneficial in COVID-19 infections given the pathophysiological processes involved in the disease. Multiple preclinical and clinical studies have shed the light on the various effects exerted by Selenium in multiple inflammatory conditions including acute lung injury and acute respiratory distress syndrome, as well as viral infections including HIV and Influenza. The study team aims to explore the possible role of Selenium in mitigating the inflammatory processes involved in COVID-19 infections and hence its effect on disease progression and mortality.

Patients with COVID-19 who exhibit the signs and symptoms of moderate or severe infection or are critically ill will receive Selenium infusion for 14 days. The working hypothesis of this trial is that selenium treatment would decrease the death rates and increase the rate of hospital discharges among hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent, or with a legal representative who can provide informed consent, or enrolled under International Conference on Harmonization (ICH) E6(R2) 4.8.15 emergency use provisions as deemed necessary by the investigator (age ≥18) prior to performing study procedure.
2. Aged ≥ 18 years.
3. Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 infection confirmed by polymerase chain reaction (PCR) test ≤ 4 days before randomization.
4. Currently hospitalized.
5. Peripheral capillary oxygen saturation (SpO2) ≤ 94% or requiring supplemental oxygen on screening.

Exclusion Criteria:

1. Participation in any other clinical trial of an experimental treatment for COVID-19.
2. Evidence of multiorgan failure.
3. Mechanically ventilated for > 5 days.
4. Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 X upper limit of normal (ULN).
5. Creatinine clearance < 50 mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Mean change in the ordinal scale | Day 1 through Day 29
  The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation; 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.
Rate of hospital discharges or deaths | Study duration
  Rate of patient discharge to home or other long-term care facilities, or death.

SECONDARY OUTCOMES:
Clinical status using ordinal scale | Day 1 through Day 29
  The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation; 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.
Mean change in the ordinal scale | Day 1 though Day 29
  The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation; 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.
Time to an improvement of one category using an ordinal scale | Day 1 though Day 29
  The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation; 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.
Change in National Early Warning Score (NEWS) from baseline | Day 1 through Day 29
  The NEW score has demonstrated an ability to discriminate patients at risk of poor outcomes. This score is based on 7 clinical parameters (respiration rate, oxygen saturation, any supplemental oxygen, temperature, systolic blood pressure, heart rate, level of consciousness). The NEW Score is being used as an efficacy measure.
Cumulative incidence of serious adverse events (SAEs) | Day 1 through Day 29
  An SAE is defined as an AE or suspected adverse reaction is considered serious if, in the view of either the investigator, it results in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
Duration of hospitalization | Day 1 though Day 29
  Measured in days.
Incidence of new oxygen use | Day 1 though Day 29
  Incidence of new oxygen use.
Duration of new oxygen use | Day 1 though Day 29
  Measured in days.
Incidence of new non-invasive ventilation or high flow oxygen use | Day 1 though Day 29
  Incidence of new non-invasive ventilation or high flow oxygen use.
Duration of new non-invasive ventilation or high flow oxygen use | Day 1 though Day 29
  Measured in days.
Incidence of new ventilator use | Day 1 though Day 29
  Incidence of new ventilator use.
Duration of new ventilator use | Day 1 though Day 29
  Measured in days.
Discontinuation or temporary suspension of investigational therapeutics | Day 1 through Day 14
  For any reason.
Change from baseline in alanine transaminase (ALT) | Day 1 through Day 29
  Change from baseline in alanine transaminase (ALT).
Change from baseline in aspartate transaminase (AST) | Day 1 through Day 29
  Change from baseline in aspartate transaminase (AST).
Change from baseline in creatinine (Cr) | Day 1 through Day 29
  Change from baseline in creatinine (Cr).
Change from baseline in glucose | Day 1 through Day 29
  Change from baseline in glucose.
Change from baseline in hemoglobin | Day 1 through Day 29
  Change from baseline in hemoglobin.
Change from baseline in platelets | Day 1 through Day 29
  Change from baseline in platelets.
Change from baseline in prothrombin time | Day 1 through Day 29
  Change from baseline in prothrombin time.
Change from baseline in total bilirubin | Day 1 through Day 29
  Change from baseline in total bilirubin.
Change from baseline in white blood cell count (WBC) with differential | Day 1 through Day 29
  Change from baseline in white blood cell count (WBC) with differential.
Change from baseline in interleukin-1 (IL-1) | Day 1 through Day 29
  Change from baseline in interleukin-1 (IL-1).
Change from baseline in interleukin-6 (IL-6) | Day 1 through Day 29
  Change from baseline in interleukin-6 (IL-6).
Change from baseline in tumor necrosis factor alpha (TNF-α) | Day 1 through Day 29
  Change from baseline in tumor necrosis factor alpha (TNF-α).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Ghoweba, MD, Principal Investigator — CHRISTUS Health
Locations (1):
- CHRISTUS Good Shepherd Medical Center, Longview, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the publication(s) after deidentification (text, tables, figures, and appendices). Proposals should be directed to mohamed.ghoweba@christushealth.org. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Perona G, Schiavon R, Guidi GC, Veneri D, Minuz P. Selenium dependent glutathione peroxidase: a physiological regulatory system for platelet function. Thromb Haemost. 1990 Oct 22;64(2):312-8. PMID 2270539
- [Background] Steinbrenner H, Sies H. Protection against reactive oxygen species by selenoproteins. Biochim Biophys Acta. 2009 Nov;1790(11):1478-85. doi: 10.1016/j.bbagen.2009.02.014. Epub 2009 Mar 5. PMID 19268692
- [Background] Steinbrenner H, Speckmann B, Klotz LO. Selenoproteins: Antioxidant selenoenzymes and beyond. Arch Biochem Biophys. 2016 Apr 1;595:113-9. doi: 10.1016/j.abb.2015.06.024. PMID 27095226
- [Background] Avery JC, Hoffmann PR. Selenium, Selenoproteins, and Immunity. Nutrients. 2018 Sep 1;10(9):1203. doi: 10.3390/nu10091203. PMID 30200430
- [Background] Hassanzadeh M, Faridhosseini R, Mahini M, Faridhosseini F, Ranjbar A. Serum Levels of TNF-, IL-6, and Selenium in Patients with Acute and Chronic Coronary Artery Disease. Iran J Immunol. 2006 Sep;3(3):142-5. doi: 10.22034/iji.2006.16988. PMID 18698124
- [Background] Zhou X, Wang Z, Chen J, Wang W, Song D, Li S, Yang H, Xue S, Chen C. Increased levels of IL-6, IL-1beta, and TNF-alpha in Kashin-Beck disease and rats induced by T-2 toxin and selenium deficiency. Rheumatol Int. 2014 Jul;34(7):995-1004. doi: 10.1007/s00296-013-2862-5. Epub 2013 Sep 15. PMID 24037056
- [Background] Gazi MH, Gong A, Donkena KV, Young CY. Sodium selenite inhibits interleukin-6-mediated androgen receptor activation in prostate cancer cells via upregulation of c-Jun. Clin Chim Acta. 2007 May 1;380(1-2):145-50. doi: 10.1016/j.cca.2007.01.031. Epub 2007 Feb 11. PMID 17346688
- [Background] Hoffmann PR, Berry MJ. The influence of selenium on immune responses. Mol Nutr Food Res. 2008 Nov;52(11):1273-80. doi: 10.1002/mnfr.200700330. PMID 18384097
- [Background] Steinbrenner H, Al-Quraishy S, Dkhil MA, Wunderlich F, Sies H. Dietary selenium in adjuvant therapy of viral and bacterial infections. Adv Nutr. 2015 Jan 15;6(1):73-82. doi: 10.3945/an.114.007575. Print 2015 Jan. PMID 25593145
- [Background] Beck MA, Levander OA, Handy J. Selenium deficiency and viral infection. J Nutr. 2003 May;133(5 Suppl 1):1463S-7S. doi: 10.1093/jn/133.5.1463S. PMID 12730444
- [Background] Beck MA. Selenium and host defence towards viruses. Proc Nutr Soc. 1999 Aug;58(3):707-11. doi: 10.1017/s0029665199000920. PMID 10604206
- [Background] Beck MA. Antioxidants and viral infections: host immune response and viral pathogenicity. J Am Coll Nutr. 2001 Oct;20(5 Suppl):384S-388S; discussion 396S-397S. doi: 10.1080/07315724.2001.10719172. PMID 11603647
- [Background] Schrauzer GN, Sacher J. Selenium in the maintenance and therapy of HIV-infected patients. Chem Biol Interact. 1994 Jun;91(2-3):199-205. doi: 10.1016/0009-2797(94)90040-x. PMID 7514960
- [Background] Hori K, Hatfield D, Maldarelli F, Lee BJ, Clouse KA. Selenium supplementation suppresses tumor necrosis factor alpha-induced human immunodeficiency virus type 1 replication in vitro. AIDS Res Hum Retroviruses. 1997 Oct 10;13(15):1325-32. doi: 10.1089/aid.1997.13.1325. PMID 9339849
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Madjid M, Safavi-Naeini P, Solomon SD, Vardeny O. Potential Effects of Coronaviruses on the Cardiovascular System: A Review. JAMA Cardiol. 2020 Jul 1;5(7):831-840. doi: 10.1001/jamacardio.2020.1286. PMID 32219363
- [Background] Wang JZ, Zhang RY, Bai J. An anti-oxidative therapy for ameliorating cardiac injuries of critically ill COVID-19-infected patients. Int J Cardiol. 2020 Aug 1;312:137-138. doi: 10.1016/j.ijcard.2020.04.009. Epub 2020 Apr 6. No abstract available. PMID 32321655
- [Background] Ahrens I, Ellwanger C, Smith BK, Bassler N, Chen YC, Neudorfer I, Ludwig A, Bode C, Peter K. Selenium supplementation induces metalloproteinase-dependent L-selectin shedding from monocytes. J Leukoc Biol. 2008 Jun;83(6):1388-95. doi: 10.1189/jlb.0707497. Epub 2008 Feb 27. PMID 18305178
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Kellner M, Noonepalle S, Lu Q, Srivastava A, Zemskov E, Black SM. ROS Signaling in the Pathogenesis of Acute Lung Injury (ALI) and Acute Respiratory Distress Syndrome (ARDS). Adv Exp Med Biol. 2017;967:105-137. doi: 10.1007/978-3-319-63245-2_8. PMID 29047084
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Vaninov N. In the eye of the COVID-19 cytokine storm. Nat Rev Immunol. 2020 May;20(5):277. doi: 10.1038/s41577-020-0305-6. No abstract available. PMID 32249847
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Zhang C, Wu Z, Li JW, Zhao H, Wang GQ. Cytokine release syndrome in severe COVID-19: interleukin-6 receptor antagonist tocilizumab may be the key to reduce mortality. Int J Antimicrob Agents. 2020 May;55(5):105954. doi: 10.1016/j.ijantimicag.2020.105954. Epub 2020 Mar 29. PMID 32234467
- [Background] Conti P, Ronconi G, Caraffa A, Gallenga CE, Ross R, Frydas I, Kritas SK. Induction of pro-inflammatory cytokines (IL-1 and IL-6) and lung inflammation by Coronavirus-19 (COVI-19 or SARS-CoV-2): anti-inflammatory strategies. J Biol Regul Homeost Agents. 2020 March-April,;34(2):327-331. doi: 10.23812/CONTI-E. PMID 32171193
- [Background] Ronco C, Reis T. Kidney involvement in COVID-19 and rationale for extracorporeal therapies. Nat Rev Nephrol. 2020 Jun;16(6):308-310. doi: 10.1038/s41581-020-0284-7. PMID 32273593
- [Background] Manzanares W, Langlois PL, Heyland DK. Pharmaconutrition with selenium in critically ill patients: what do we know? Nutr Clin Pract. 2015 Feb;30(1):34-43. doi: 10.1177/0884533614561794. Epub 2014 Dec 18. PMID 25524883
- [Background] Angstwurm MW, Engelmann L, Zimmermann T, Lehmann C, Spes CH, Abel P, Strauss R, Meier-Hellmann A, Insel R, Radke J, Schuttler J, Gartner R. Selenium in Intensive Care (SIC): results of a prospective randomized, placebo-controlled, multiple-center study in patients with severe systemic inflammatory response syndrome, sepsis, and septic shock. Crit Care Med. 2007 Jan;35(1):118-26. doi: 10.1097/01.CCM.0000251124.83436.0E. PMID 17095947
- [Background] Heyland DK, Dhaliwal R, Suchner U, Berger MM. Antioxidant nutrients: a systematic review of trace elements and vitamins in the critically ill patient. Intensive Care Med. 2005 Mar;31(3):327-37. doi: 10.1007/s00134-004-2522-z. Epub 2004 Dec 17. PMID 15605227
- [Background] Hardy G, Hardy I, Manzanares W. Selenium supplementation in the critically ill. Nutr Clin Pract. 2012 Feb;27(1):21-33. doi: 10.1177/0884533611434116. PMID 22307489
- [Background] Allingstrup M, Afshari A. Selenium supplementation for critically ill adults. Cochrane Database Syst Rev. 2015 Jul 27;2015(7):CD003703. doi: 10.1002/14651858.CD003703.pub3. PMID 26214143
- [Background] Schmidt T, Pargger H, Seeberger E, Eckhart F, von Felten S, Haberthur C. Effect of high-dose sodium selenite in cardiac surgery patients: A randomized controlled bi-center trial. Clin Nutr. 2018 Aug;37(4):1172-1180. doi: 10.1016/j.clnu.2017.04.019. Epub 2017 May 2. PMID 28502744
- [Background] Bargagli E, Olivieri C, Bennett D, Prasse A, Muller-Quernheim J, Rottoli P. Oxidative stress in the pathogenesis of diffuse lung diseases: a review. Respir Med. 2009 Sep;103(9):1245-56. doi: 10.1016/j.rmed.2009.04.014. Epub 2009 May 22. PMID 19464864
- [Background] Ghosh P, Bhattacharjee A, Basu A, Singha Roy S, Bhattacharya S. Attenuation of cyclophosphamide-induced pulmonary toxicity in Swiss albino mice by naphthalimide-based organoselenium compound 2-(5-selenocyanatopentyl)-benzo[de]isoquinoline 1,3-dione. Pharm Biol. 2015 Apr;53(4):524-32. doi: 10.3109/13880209.2014.931440. Epub 2014 Dec 4. PMID 25471377
- [Background] Kim KS, Suh GJ, Kwon WY, Kwak YH, Lee K, Lee HJ, Jeong KY, Lee MW. Antioxidant effects of selenium on lung injury in paraquat intoxicated rats. Clin Toxicol (Phila). 2012 Sep;50(8):749-53. doi: 10.3109/15563650.2012.708418. PMID 22924652
- [Background] Liu J, Yang Y, Zeng X, Bo L, Jiang S, Du X, Xie Y, Jiang R, Zhao J, Song W. Investigation of selenium pretreatment in the attenuation of lung injury in rats induced by fine particulate matters. Environ Sci Pollut Res Int. 2017 Feb;24(4):4008-4017. doi: 10.1007/s11356-016-8173-0. Epub 2016 Dec 5. PMID 27921246
- [Background] Amini P, Kolivand S, Saffar H, Rezapoor S, Motevaseli E, Najafi M, Nouruzi F, Shabeeb D, Musa AE. Protective Effect of Selenium-L-methionine on Radiation-induced Acute Pneumonitis and Lung Fibrosis in Rat. Curr Clin Pharmacol. 2019;14(2):157-164. doi: 10.2174/1574884714666181214101917. PMID 30556505
- [Background] Zhang Y, Jiang M, Nouraie M, Roth MG, Tabib T, Winters S, Chen X, Sembrat J, Chu Y, Cardenes N, Tuder RM, Herzog EL, Ryu C, Rojas M, Lafyatis R, Gibson KF, McDyer JF, Kass DJ, Alder JK. GDF15 is an epithelial-derived biomarker of idiopathic pulmonary fibrosis. Am J Physiol Lung Cell Mol Physiol. 2019 Oct 1;317(4):L510-L521. doi: 10.1152/ajplung.00062.2019. Epub 2019 Aug 21. PMID 31432710
- [Background] Kempf T, Wollert KC. Risk stratification in critically ill patients: GDF-15 scores in adult respiratory distress syndrome. Crit Care. 2013 Jul 31;17(4):173. doi: 10.1186/cc12765. PMID 23905849
- [Background] Jaspers I, Zhang W, Brighton LE, Carson JL, Styblo M, Beck MA. Selenium deficiency alters epithelial cell morphology and responses to influenza. Free Radic Biol Med. 2007 Jun 15;42(12):1826-37. doi: 10.1016/j.freeradbiomed.2007.03.017. Epub 2007 Mar 24. PMID 17512462
- [Background] Tindell R, Wall SB, Li Q, Li R, Dunigan K, Wood R, Tipple TE. Selenium supplementation of lung epithelial cells enhances nuclear factor E2-related factor 2 (Nrf2) activation following thioredoxin reductase inhibition. Redox Biol. 2018 Oct;19:331-338. doi: 10.1016/j.redox.2018.07.020. Epub 2018 Sep 5. PMID 30212802
- [Background] Rojo de la Vega M, Dodson M, Gross C, Mansour HM, Lantz RC, Chapman E, Wang T, Black SM, Garcia JG, Zhang DD. Role of Nrf2 and Autophagy in Acute Lung Injury. Curr Pharmacol Rep. 2016 Apr;2(2):91-101. doi: 10.1007/s40495-016-0053-2. Epub 2016 Feb 6. PMID 27313980
- [Background] Zhang C, Lin J, Ge J, Wang LL, Li N, Sun XT, Cao HB, Li JL. Selenium triggers Nrf2-mediated protection against cadmium-induced chicken hepatocyte autophagy and apoptosis. Toxicol In Vitro. 2017 Oct;44:349-356. doi: 10.1016/j.tiv.2017.07.027. Epub 2017 Jul 29. PMID 28765097
- [Background] Sakr Y, Reinhart K, Bloos F, Marx G, Russwurm S, Bauer M, Brunkhorst F. Time course and relationship between plasma selenium concentrations, systemic inflammatory response, sepsis, and multiorgan failure. Br J Anaesth. 2007 Jun;98(6):775-84. doi: 10.1093/bja/aem091. Epub 2007 May 3. PMID 17478454
- [Background] Ricetti MM, Guidi GC, Bellisola G, Marrocchella R, Rigo A, Perona G. Selenium enhances glutathione peroxidase activity and prostacyclin release in cultured human endothelial cells. Concurrent effects on mRNA levels. Biol Trace Elem Res. 1994 Oct-Nov;46(1-2):113-23. doi: 10.1007/BF02790072. PMID 7888276
- [Background] Fontaine M, Valli VE, Young LG. Studies on vitamin E and selenium deficiency in young pigs. IV. Effect on coagulation system. Can J Comp Med. 1977 Jan;41(1):64-76. PMID 832191
- [Background] Zhang Y, Xiao M, Zhang S, Xia P, Cao W, Jiang W, Chen H, Ding X, Zhao H, Zhang H, Wang C, Zhao J, Sun X, Tian R, Wu W, Wu D, Ma J, Chen Y, Zhang D, Xie J, Yan X, Zhou X, Liu Z, Wang J, Du B, Qin Y, Gao P, Qin X, Xu Y, Zhang W, Li T, Zhang F, Zhao Y, Li Y, Zhang S. Coagulopathy and Antiphospholipid Antibodies in Patients with Covid-19. N Engl J Med. 2020 Apr 23;382(17):e38. doi: 10.1056/NEJMc2007575. Epub 2020 Apr 8. PMID 32268022
- [Background] Ma X, Bi S, Wang Y, Chi X, Hu S. Combined adjuvant effect of ginseng stem-leaf saponins and selenium on immune responses to a live bivalent vaccine of Newcastle disease virus and infectious bronchitis virus in chickens. Poult Sci. 2019 Sep 1;98(9):3548-3556. doi: 10.3382/ps/pez207. PMID 31220864
- [Background] Marty AM, Jones MK. The novel Coronavirus (SARS-CoV-2) is a one health issue. One Health. 2020 Feb 14;9:100123. doi: 10.1016/j.onehlt.2020.100123. eCollection 2020 Jun. No abstract available. PMID 32140538
- [Background] Chu VC, McElroy LJ, Chu V, Bauman BE, Whittaker GR. The avian coronavirus infectious bronchitis virus undergoes direct low-pH-dependent fusion activation during entry into host cells. J Virol. 2006 Apr;80(7):3180-8. doi: 10.1128/JVI.80.7.3180-3188.2006. PMID 16537586
- [Background] Weiss SR, Navas-Martin S. Coronavirus pathogenesis and the emerging pathogen severe acute respiratory syndrome coronavirus. Microbiol Mol Biol Rev. 2005 Dec;69(4):635-64. doi: 10.1128/MMBR.69.4.635-664.2005. PMID 16339739
- [Background] Wu C, Liu Y, Yang Y, Zhang P, Zhong W, Wang Y, Wang Q, Xu Y, Li M, Li X, Zheng M, Chen L, Li H. Analysis of therapeutic targets for SARS-CoV-2 and discovery of potential drugs by computational methods. Acta Pharm Sin B. 2020 May;10(5):766-788. doi: 10.1016/j.apsb.2020.02.008. Epub 2020 Feb 27. PMID 32292689
- [Background] Zhang J, Taylor EW, Bennett K, Saad R, Rayman MP. Association between regional selenium status and reported outcome of COVID-19 cases in China. Am J Clin Nutr. 2020 Jun 1;111(6):1297-1299. doi: 10.1093/ajcn/nqaa095. No abstract available. PMID 32342979
- [Background] Zhao Y, Yang M, Mao Z, Yuan R, Wang L, Hu X, Zhou F, Kang H. The clinical outcomes of selenium supplementation on critically ill patients: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2019 May;98(20):e15473. doi: 10.1097/MD.0000000000015473. PMID 31096444
- [Background] Angstwurm MW, Gaertner R. Practicalities of selenium supplementation in critically ill patients. Curr Opin Clin Nutr Metab Care. 2006 May;9(3):233-8. doi: 10.1097/01.mco.0000222105.30795.7f. PMID 16607122
- [Background] Manzanares W, Biestro A, Galusso F, Torre MH, Manay N, Facchin G, Hardy G. High-dose selenium for critically ill patients with systemic inflammation: pharmacokinetics and pharmacodynamics of selenious acid: a pilot study. Nutrition. 2010 Jun;26(6):634-40. doi: 10.1016/j.nut.2009.06.022. Epub 2010 Jan 15. PMID 20080034
- [Background] Nuttall KL. Evaluating selenium poisoning. Ann Clin Lab Sci. 2006 Autumn;36(4):409-20. PMID 17127727